CLINICAL TRIAL: NCT07324135
Title: A Double-blind Randomized Controlled Study to Evaluate the Effect of Young Child Formula on Iron Status in Children 1-3 Years of Age.
Brief Title: Effect of Young Child Formula on Iron Status in Children 1-3 Years of Age.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 24REX0077885
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Iron Status
Keywords: YCF; Young Child Formula; Anaemia; Iron status
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, parallel-group, multi-centre intervention study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product (Experimental): Young Child Formula
  Interventions: Other: Nutritional product
- Control product (Other): Control: cow's milk
  Interventions: Other: Nutritional product

INTERVENTIONS:
Other: Nutritional product — parents will be instructed to provide subjects with 2-3 servings of Study Product per day

SUMMARY:
This study evaluates the effect of young child formula in children 1-3 years of age. Subjects will receive either test or control product. Growth and health data, parent diaries and biological samples will be collected during the study.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 3 years
* Healthy children (as per investigator clinical judgement and non-anaemic as confirmed by Hb levels) or meeting the criteria for mild anaemia based on Hb levels
* Children familiar with drinking milk products (in combination with breastfeeding or not) for at least 3 weeks prior to screening.
* Written informed consent provided by parent(s) / legally acceptable representative(s) aged ≥18 years at screening

Exclusion Criteria:

* Low Hb meeting the criteria for moderate or severe anaemia
* Use of iron and/or fibre supplementation within 3 months prior to screening
* Any infection within 2 weeks prior to screening
* Any other medical condition with known high CRP (>5 mg/L) / high AGP (>1 g/L) value within 2 weeks prior to screening
* The use of medication that is likely to interfere with iron metabolism) within 2 weeks prior to screening
* The use of medication to treat iron deficiency or anaemia within 3 months prior to screening
* Any developmental delays that could impact feeding behaviour or growth, or any other condition that is likely to influence nutritional status or growth.
* Disorders requiring a special diet.
* Any other iron metabolism and related disorders
* Children with known or suspected medical conditions requiring a special diet or special formulae, food allergy, or food intolerances.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 466 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Serum ferritin concentration | Baseline and 20 weeks post baseline

SECONDARY OUTCOMES:
Daily iron intake | Baseline, 10 weeks and 20 weeks post-baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine University of Indonesia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No